CLINICAL TRIAL: NCT03899155
Title: Pan-Tumor Study for Long-term Treatment of Cancer Patients Who Have Participated in BMS Sponsored Trials Investigating Nivolumab and Other Cancer Therapies
Brief Title: Pan Tumor Rollover Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Exelixis (Industry); Novartis (Industry); Clovis Oncology, Inc. (Industry); Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-8TT; 2018-004362-34 (EudraCT Number)
Record Dates: First submitted 2019-04-01; First posted 2019-04-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cancer
Keywords: Rollover; pan-tumor
MeSH Terms: conditions — Neoplasms | interventions — Nivolumab; Ipilimumab; cabozantinib; trametinib; relatlimab; Capecitabine; Bevacizumab; Temozolomide; rucaparib; daratumumab; Leucovorin; Fluorouracil; Oxaliplatin; enzalutamide; Sunitinib; Pemetrexed; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (32):
- A1: Nivolumab Monotherapy Dose 1 (Experimental)
  Interventions: Drug: Nivolumab
- A2: Nivolumab Monotherapy Dose 2 (Experimental)
  Interventions: Drug: Nivolumab
- B1: Nivolumab + Ipilimumab (Experimental)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- B2: Nivolumab + Ipilimumab + Cabozantinib (Experimental)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Cabozantinib
- B3: Nivolumab + Ipilimumab + Trametinib (Experimental)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Trametinib
- C1: Relatlimab + Nivolumab Fixed Dose Combination Dose 1 (Experimental)
  Interventions: Drug: Nivolumab + Relatlimab
- C3: Relatlimab + Nivolumab Fixed Dose Combination Dose 2 (Experimental)
  Interventions: Drug: Nivolumab + Relatlimab
- C2: Relatlimab + Nivolumab Single Agent Vial (SAV) Dose 1 (Experimental)
  Interventions: Drug: Nivolumab; Drug: Relatlimab
- C4: Relatlimab + Nivolumab SAV Dose 2 (Experimental)
  Interventions: Drug: Nivolumab; Drug: Relatlimab
- C5: Relatlimab + Nivolumab + Ipilimumab (Experimental)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- C6: Relatlimab + Nivolumab + Capecitabine (Experimental)
  Interventions: Drug: Nivolumab + Relatlimab; Drug: Capecitabine
- C7: Relatlimab + Nivolumab SAV Dose 3 (Experimental)
  Interventions: Drug: Nivolumab; Drug: Relatlimab
- C10: Relatlimab + Nivolumab SAV Dose 4 (Experimental)
  Interventions: Drug: Nivolumab; Drug: Relatlimab
- C12: Relatlimab + Nivolumab SAV Dose 5 (Experimental)
  Interventions: Drug: Nivolumab; Drug: Relatlimab
- C8: Relatlimab + Nivolumab SAV + PDCT Dose 1 (Experimental)
  Interventions: Drug: Nivolumab; Drug: Relatlimab
- C9: Relatlimab + Nivolumab SAV + Bevacizumab (Experimental)
  Interventions: Drug: Nivolumab; Drug: Relatlimab; Drug: Bevacizumab
- C11: Relatlimab + Nivolumab SAV + PDCT Dose 2 (Experimental)
  Interventions: Drug: Nivolumab; Drug: Relatlimab
- D1: Nivolumab + Temozolomide (Experimental)
  Interventions: Drug: Nivolumab; Drug: Temozolomide
- D2: Nivolumab + Rucaparib (Experimental)
  Interventions: Drug: Nivolumab; Drug: Rucaparib
- D3: Nivolumab + Daratumumab (Experimental)
  Interventions: Drug: Nivolumab; Drug: Daratumumab
- D4: Nivolumab + Bevacizumab (Experimental)
  Interventions: Drug: Nivolumab
- E1: Bevacizumab Monotherapy (Experimental)
  Interventions: Drug: Bevacizumab
- E2: Regorafinib Monotherapy (Experimental)
  Interventions: Drug: Regorafinib
- E4: Leucovorin + Oxaliplatin + Fluorouracil (Experimental)
  Interventions: Drug: Leucovorin; Drug: Fluorouracil; Drug: Oxaliplatin
- E5: Enzalutamide Monotherapy (Experimental)
  Interventions: Drug: Enzalutamide
- E6: Sunitinib Monotherapy (Experimental)
  Interventions: Drug: Sunitinib
- E7: Rucaparib Monotherapy (Experimental)
  Interventions: Drug: Rucaparib
- E8: Capecitabine Monotherapy (Experimental)
  Interventions: Drug: Capecitabine
- E9: Cabozantinib Monotherapy (Experimental)
  Interventions: Drug: Cabozantinib
- E10: Pemetrexed Monotherapy (Experimental)
  Interventions: Drug: Pemetrexed
- E11: Pembrolizumab Monotherapy (Experimental)
  Interventions: Drug: Pembrolizumab
- E3: Leucovorin + Fluorouracil (Experimental)
  Interventions: Drug: Leucovorin

INTERVENTIONS:
Drug: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558-01
  Arms: A1: Nivolumab Monotherapy Dose 1; A2: Nivolumab Monotherapy Dose 2; B1: Nivolumab + Ipilimumab; B2: Nivolumab + Ipilimumab + Cabozantinib; B3: Nivolumab + Ipilimumab + Trametinib; C10: Relatlimab + Nivolumab SAV Dose 4; C11: Relatlimab + Nivolumab SAV + PDCT Dose 2; C12: Relatlimab + Nivolumab SAV Dose 5; C2: Relatlimab + Nivolumab Single Agent Vial (SAV) Dose 1; C4: Relatlimab + Nivolumab SAV Dose 2; C5: Relatlimab + Nivolumab + Ipilimumab; C7: Relatlimab + Nivolumab SAV Dose 3; C8: Relatlimab + Nivolumab SAV + PDCT Dose 1; C9: Relatlimab + Nivolumab SAV + Bevacizumab; D1: Nivolumab + Temozolomide; D2: Nivolumab + Rucaparib; D3: Nivolumab + Daratumumab; D4: Nivolumab + Bevacizumab
Drug: Ipilimumab — Specified dose on specified days
  Arms: B1: Nivolumab + Ipilimumab; B2: Nivolumab + Ipilimumab + Cabozantinib; B3: Nivolumab + Ipilimumab + Trametinib; C5: Relatlimab + Nivolumab + Ipilimumab
Drug: Cabozantinib — Specified dose on specified days
  Arms: B2: Nivolumab + Ipilimumab + Cabozantinib; E9: Cabozantinib Monotherapy
Drug: Trametinib — Specified dose on specified days
  Arms: B3: Nivolumab + Ipilimumab + Trametinib
Drug: Relatlimab — Specified dose on specified days
  Other Names: BMS-986016-01
  Arms: C10: Relatlimab + Nivolumab SAV Dose 4; C11: Relatlimab + Nivolumab SAV + PDCT Dose 2; C12: Relatlimab + Nivolumab SAV Dose 5; C2: Relatlimab + Nivolumab Single Agent Vial (SAV) Dose 1; C4: Relatlimab + Nivolumab SAV Dose 2; C7: Relatlimab + Nivolumab SAV Dose 3; C8: Relatlimab + Nivolumab SAV + PDCT Dose 1; C9: Relatlimab + Nivolumab SAV + Bevacizumab
Drug: Nivolumab + Relatlimab — Specified dose on specified days
  Other Names: BMS-986213
  Arms: C1: Relatlimab + Nivolumab Fixed Dose Combination Dose 1; C3: Relatlimab + Nivolumab Fixed Dose Combination Dose 2; C6: Relatlimab + Nivolumab + Capecitabine
Drug: Capecitabine — Specified dose on specified days
  Arms: C6: Relatlimab + Nivolumab + Capecitabine; E8: Capecitabine Monotherapy
Drug: Bevacizumab — Specified dose on specified days
  Arms: C9: Relatlimab + Nivolumab SAV + Bevacizumab; E1: Bevacizumab Monotherapy
Drug: Temozolomide — Specified dose on specified days
  Arms: D1: Nivolumab + Temozolomide
Drug: Rucaparib — Specified dose on specified days
  Arms: D2: Nivolumab + Rucaparib; E7: Rucaparib Monotherapy
Drug: Daratumumab — Specified dose on specified days
  Arms: D3: Nivolumab + Daratumumab
Drug: Regorafinib — Specified dose on specified days
  Arms: E2: Regorafinib Monotherapy
Drug: Leucovorin — Specified dose on specified days
  Arms: E3: Leucovorin + Fluorouracil; E4: Leucovorin + Oxaliplatin + Fluorouracil
Drug: Fluorouracil — Specified dose on specified days
  Arms: E4: Leucovorin + Oxaliplatin + Fluorouracil
Drug: Oxaliplatin — Specified dose on specified days
  Arms: E4: Leucovorin + Oxaliplatin + Fluorouracil
Drug: Enzalutamide — Specified dose on specified days
  Arms: E5: Enzalutamide Monotherapy
Drug: Sunitinib — Specified dose on specified days
  Arms: E6: Sunitinib Monotherapy
Drug: Pemetrexed — Specified dose on specified days
  Arms: E10: Pemetrexed Monotherapy
Drug: Pembrolizumab — Specified dose on specified days
  Arms: E11: Pembrolizumab Monotherapy

SUMMARY:
Main Objective of this study is to examine long-term safety of nivolumab monotherapy including combinations and other cancer therapies in various tumor types.

ELIGIBILITY:
Inclusion Criteria

* Signed Written Informed Consent.
* Eligible to receive continued study treatment per the Parent Study, including treatment beyond progression per investigator assessment in the Parent Study.
* On treatment hold in the Parent Study following long-lasting response or are eligible for treatment rechallenge as defined in the Parent Study.
* WOCBP and male participants who are sexually active must agree to follow instructions for method(s) of contraception as described below and included in the ICF.

Exclusion Criteria

* Participant is not eligible for study treatment per the Parent Study eligibility criteria.
* Participants not receiving clinical benefit as assessed by the Investigator.
* Any clinical adverse event (AE), laboratory abnormality, or intercurrent illness which, in the opinion of the Investigator, indicates that participation in the study is not in the best interest of the participant.
* Other protocol-defined Inclusion/Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2029-08-25 (Estimated); Study Completion 2029-08-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | From Day 1 up to 135 Days after discontinuation of treatment
Incidence of drug related AEs | From Day 1 up to 135 Days after discontinuation of treatment
Incidence of AEs leading to Discontinuation | From Day 1 up to 135 Days after discontinuation of treatment
Incidence of Serious Adverse Events (SAEs) | From signature of Informed Consent up to 135 Days after discontinuation of treatment
Incidence of Select AEs | From Day 1 up to 135 Days after discontinuation of treatment
Incidence of Immune-Mediated AEs | From Day 1 up to 135 Days after discontinuation of treatment
Incidence of Death | From signature of Informed Consent up to 135 Days after discontinuation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (395):
- United States (58):
  - Local Institution - 0220, Huntsville, Alabama
  - University of Arizona College of Medicine, Tucson, Arizona
  - Innovative Clinical Research Institute, Lynwood, California
  - Local Institution, San Francisco, California
  - Local Institution - 0099, San Francisco, California
  - Local Institution - 0233, Aurora, Colorado
  - Local Institution - 0095, New Haven, Connecticut
  - Local Institution - 0088, Washington D.C., District of Columbia
  - Florida Cancer Affiliates, Ocala, Florida
  - Local Institution, Orlando, Florida
  - Local Institution - 0024, Tampa, Florida
  - Local Institution - 0105, Chicago, Illinois
  - Local Institution, Maywood, Illinois
  - Local Institution - 0279, Park Ridge, Illinois
  - Local Institution - 0186, Westwood, Kansas
  - Local Institution - 0165, Wichita, Kansas
  - University of Louisville-James Graham Brown Cancer Center, Louisville, Kentucky
  - Local Institution - 0092, Baltimore, Maryland
  - Local Institution - 0039, Boston, Massachusetts
  - Dana_Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Local Institution - 0081, Boston, Massachusetts
  - Local Institution - 0143, Ann Arbor, Michigan
  - Local Institution - 0100, Minneapolis, Minnesota
  - Local Institution, St Louis, Missouri
  - Local Institution - 0205, Omaha, Nebraska
  - Local Institution - 0014, Lebanon, New Hampshire
  - Local Institution, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hematology Oncology Associates-Mineola, Mineola, New York
  - Local Institution, New York, New York
  - Local Institution - 0185, New York, New York
  - Local Institution - 0202, New York, New York
  - Local Institution - 0204, Charlotte, North Carolina
  - Local Institution - 0016, Durham, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
  - Local Institution, Cleveland, Ohio
  - The Ohio University, Columbus, Ohio
  - Local Institution - 0246, Tulsa, Oklahoma
  - Local Institution - 0037, Allentown, Pennsylvania
  - Local Institution - 0054, Easton, Pennsylvania
  - Lancaster General Health, Lancaster, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution - 0162, Philadelphia, Pennsylvania
  - Local Institution - 0110, Pittsburgh, Pennsylvania
  - Local Institution - 0228, Charleston, South Carolina
  - Local Institution, Greenville, South Carolina
  - Local Institution, Chattanooga, Tennessee
  - Tennesse Oncology, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Local Institution, Dallas, Texas
  - Local Institution - 0364, Houston, Texas
  - Local Institution - 0055, Salt Lake City, Utah
  - Local Institution, Charlottesville, Virginia
  - Public Hospital of King County District 1 Valley Medical Center, Renton, Washington
  - Local Institution - 0065, Madison, Wisconsin
  - Local Institution - 0124, Madison, Wisconsin
- Argentina (11):
  - Local Institution - 0199, Berazategui, Buenos Aires
  - Instituto Medico Rio Cuarto, Río Cuarto, Córdoba Province
  - Centro de Investigaciones Clinicas. Clinica Viedma S.A., Viedma, Río Negro Province
  - Sanatorio Parque, Rosario, Santa Fe Province
  - CAIPO Centro para la Atencion Integral del Paciente Oncologico, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0191, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0201, Buenos Aires
  - Instituto Fleming, Buenos Aires
  - Local Institution, CABA
  - Fundacion Richardet Longo - IONC, Córdoba
  - Local Institution - 0170, Córdoba
- Australia (15):
  - Local Institution - 0045, Coffs Harbour, New South Wales
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Chris OBrien Lifehouse Hospital, Sydney, New South Wales
  - Local Institution - 0193, Waratah, New South Wales
  - Local Institution - 0208, Westmead, New South Wales
  - Gallipoli Medical Foundation, Greenslopes, Queensland
  - Local Institution - 0372, Greenslopes, Queensland
  - Local Institution, South Brisbane, Queensland
  - Tasman Oncology Research Ltd, Southport, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution - 0196, Elizabeth Vale, South Australia
  - BRICC - Ballarat Health Services, Ballarat, Victoria
  - Local Institution - 0365, Fitzroy, Victoria
  - Cabrini Hospital Malvern, Malvern, Victoria
  - Local Institution - 0174, Murdoch, Western Australia
- Austria (5):
  - Local Institution - 0254, Graz, Styria
  - Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria
  - Allgemeines Krankenhaus Wien, Vienna
  - Local Institution - 0104, Vienna
  - Local Institution - 0145, Wels
- Belgium (6):
  - Local Institution - 0329, Brussels
  - Local Institution - 0232, Ghent
  - Local Institution - 0139, Jette
  - Local Institution - 0261, Liège
  - Local Institution - 0293, Sint-Niklaas
  - Local Institution - 0157, Yvoir
- Brazil (15):
  - Local Institution - 0260, Belo Horizonte, Minas Gerais
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia, Ijuí, Rio Grande do Sul
  - Local Institution - 0379, Passo Fundo, Rio Grande do Sul
  - Local Institution - 0093, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas Da Pucrs, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0399, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0264, Barretos, São Paulo
  - Local Institution - 0262, São José do Rio Preto, São Paulo
  - ICESP - Instituto do Cancer do Estado de Soo Paulo, São Paulo, São Paulo
  - Local Institution - 0263, São Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
  - Local Institution - 0266, Rio de Janeiro
  - Local Institution - 0258, Rio de Janeiro
  - Local Institution - 0340, São Paulo
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Halifax, Nova Scotia
  - Local Institution - 0168, Oshawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Local Institution - 0040, Montreal, Quebec
  - Local Institution - 0308, Montreal, Quebec
- Chile (6):
  - Local Institution - 0363, Temuco, Región de la Araucanía
  - Orlandi Oncologia, Providencia, Santiago Metropolitan
  - Bradford Hill Centro de Investigacion Clinica, Santiago, Santiago Metropolitan
  - Fundacion Arturo Lopez Perez, Santiago, Santiago Metropolitan
  - Local Institution, Santiago, Santiago Metropolitan
  - Local Institution - 0079, Viña del Mar
- China (23):
  - Local Institution - 0169, Hefei, Anhui
  - Local Institution - 0198, Beijing, Beijing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Nanfang Hospital; Southern Medical University, Guangzhou, Guangdong
  - Local Institution - 0245, Harbin, Heilongjiang
  - Harbin Medical University - Cancer Hospital, Harbin, Heilongjiang
  - Local Institution - 0160, Harbin, Heilongjiang
  - Local Institution - 0172, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Local Institution - 0348, Nanjing, Jiangsu
  - Jilin University (JLU) - First Affiliated Hospital - Cancer Center, Changchun, Jilin
  - Jilin Cancer Hospital, Changchun, Jilin
  - Tangdu Hospital of Fourth Military Medical University, Xi'an, Shaanxi
  - Xian International Medical Center Hospital, Xi'an, Shan3XI
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Fudan University - Shanghai Cancer Center FUSCC, Shanghai, Shanghai Municipality
  - Local Institution - 0278, Shanghai, Shanghai Municipality
  - Local Institution - 0325, Shanghai, Shanghai Municipality
  - Local Institution - 0188, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital Zhejiang University (The First Hospital of Zhejiang Province), Hangzhou
  - Jiangsu Cancer Hospital, Nanjing
- Czechia (5):
  - Local Institution - 0371, Brno
  - FNHK Klinika onkologie a radioterapie, Hradec Králové
  - Local Institution - 0150, Olomouc
  - Local Institution - 0253, Prague
  - Local Institution - 0275, Prague
- Local Institution, Odense C, Denmark
- Local Institution, Helsinki, Finland
- France (25):
  - Local Institution - 0006, Bordeaux, Gironde
  - CHU De Nancy Hopital De Brabois, Vandœuvre-lès-Nancy, Meurthe-Et-Moselle
  - Centre Jean Perrin, Clermont-Ferrand
  - Local Institution - 0107, Créteil
  - Local Institution - 0074, Dijon
  - Local Institution - 0109, Dijon
  - CHU Grenobles Alpes, La Tronche
  - Pole Biologie Pathologie Genetique - CHU de Lille, Lille
  - APHM - Hopital de la Timone, Marseille
  - Local Institution - 0153, Marseille
  - CHU Montpellier, Montpellier
  - Local Institution, Montpellier
  - CHU Nantes - Hotel Dieu, Nantes
  - Local Institution - 0300, Nantes
  - Local Institution - 0028, Paris
  - Local Institution - 0301, Paris
  - Local Institution - 0167, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Local Institution, Rennes
  - CHU de Saint-Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - Hopital Foch, Suresnes
  - Local Institution - 0156, Toulon
  - Local Institution, Toulouse
  - Institut Gustave Roussy, Villejuif
  - Local Institution - 0387, Paris, Île-de-France Region
- Germany (31):
  - Local Institution - 0386, Löwenstein, Baden-Wurttemberg
  - Local Institution - 0276, Munich, Bavaria
  - Local Institution - 0332, Nuremberg, Bavaria
  - Evangelische Kliniken Essen Mitte. Evang. Huyssens-Stiftung Essen-Huttrop, Essen, North Rhine-Westphalia
  - Local Institution - 0250, Essen, North Rhine-Westphalia
  - Local Institution - 0375, Essen, North Rhine-Westphalia
  - Universitaetsklinikum Aachen, Aachen
  - Local Institution - 0248, Berlin
  - Local Institution - 0249, Buxtehude
  - Local Institution - 0296, Cologne
  - Local Institution, Cologne
  - University of Freiburg, Freiburg im Breisgau
  - Local Institution, Gera
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Local Institution - 0076, Göttingen
  - Local Institution, Göttingen
  - Local Institution - 0241, Hamburg
  - Local Institution, Heidelberg
  - Thoraxklinik, Heidelberg
  - Local Institution - 0342, Heidelberg
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Universitaetsklinikum Jena - Klinik und Poliklinik fuer Urologie, Jena
  - Local Institution - 0288, Kassel
  - Local Institution - 0072, Kiel
  - Local Institution, Kiel
  - Local Institution - 0298, Löwenstein
  - Local Institution - 0098, Lübeck
  - Local Institution - 0089, Mainz
  - Local Institution, Mainz
  - Local Institution - 0017, Tübingen
  - Local Institution - 0277, Tübingen
- Greece (9):
  - Alexandra Hospital, Athens, Attica
  - Local Institution - 0244, Heraklion, Crete
  - General Hospital of Athens Laiko, Athens
  - Local Institution - 0126, Athens
  - Local Institution - 0171, Athens
  - Local Institution - 0042, Athens
  - Local Institution - 0295, Athens
  - Local Institution, Pátrai
  - Local Institution - 0215, Thessaloniki
- Queen Mary Hospital, Hong Kong, Hong Kong
- Hungary (4):
  - Local Institution - 0290, Gyöngyössolymos, Heves County
  - Local Institution - 0159, Budapest
  - Local Institution - 0226, Budapest
  - Local Institution - 0187, Debrecen
- Ireland (2):
  - Local Institution - 0227, Dublin
  - Local Institution, Limerick
- Israel (5):
  - Local Institution - 0190, Haifa
  - Local Institution - 0270, Jerusalem
  - Local Institution, Petah Tikva
  - Local Institution - 0052, Ramat Gan
  - Local Institution - 0350, Tiqwa
- Italy (26):
  - IRCCS - Istituto Scientifico Romagnolo per lo Studio dei Tumori - Dino Amadori - Srl, Meldola, Fc
  - Local Institution - 0333, Rozzano, MI
  - Istituto Nazionale dei Tumori Regina Elena, Roma, RM
  - Local Institution - 0034, Bari
  - ASST Papa Giovanni XXIII - Unita di Oncologia, Bergamo
  - Local Institution - 0326, Candiolo
  - "Azienda Ospedaliero - Universitaria ""Policlinico-Vittorio Emanuele"" - Ospedale Gaspare Rodolico", Catania
  - Local Institution - 0251, Genova
  - Local Institution, Genova
  - Local Institution - 0108, Meldola
  - Local Institution - 0303, Meldola
  - Fondazione IRCCS istituto Neurologico Carlo Besta;, Milan
  - Local Institution - 0096, Milan
  - Local Institution - 0351, Milan
  - Local Institution, Milan
  - Local Institution - 0071, Milan
  - Local Institution - 0267, Milan
  - Local Institution - 0327, Modena
  - Istituto Nazionale Tumori - Fondazione Pascale Italy, Napoli
  - Local Institution - 0218, Napoli
  - Local Institution - 0292, Napoli
  - Istituto Oncologico Veneto, Padua
  - Local Institution - 0180, Ravenna
  - Local Institution - 0003, Siena
  - Local Institution - 0291, Terni
  - Azienda Ospedaliera Citta della Salute e della Scienza, Torino
- Japan (23):
  - Local Institution - 0242, Hirosaki-shi, Aomori
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa-Shi, Chiba
  - Ehime Prefectural Central Hospital, Matsuyama, Ehime
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Local Institution - 0211, Kobe, Hyōgo
  - Local Institution - 0240, Tsukuba, Ibaraki
  - Local Institution - 0219, Kanazawa, Ishikawa-ken
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Local Institution - 0222, Natori-shi, Miyagi
  - Local Institution - 0230, Niigata, Niigata
  - Local Institution - 0214, Sayama, Osaka
  - Local Institution - 0212, Takatsuki, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Tokyo Women's Medical University - Adachi Medical Center, Adachi-Ku, Tokyo
  - Institute of Science Tokyo Hospital, Bunkyo-Ku, Tokyo
  - Local Institution - 0235, Chuo-ku, Tokyo
  - Local Institution - 0217, Koto-Ku, Tokyo
  - Local Institution - 0239, Shinjuku, Tokyo
  - Local Institution - 0224, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Local Institution - 0236, Niigata
- Mexico (14):
  - Local Institution - 0152, León, Guanajuato
  - Investigación Biomédica para el Desarrollo de Fármacos S.A de C.V, Zapopan, Jalisco
  - Cryptex Investigacion Clinica Sa de Cv, Cuauhtémoc, Mexico City
  - Local Institution - 0181, Tlalpan, Mexico City
  - Local Institution - 0007, Morelia, Michoacán
  - Local Institution - 0286, Monterrey, Nuevo León
  - Local Institution - 0354, Monterrey, Nuevo León
  - I Can Oncology Center, Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City, Oaxaca
  - Local Institution - 0343, Querétaro City, Querétaro
  - Local Institution - 0410, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - Instituto Nacional de Cancerologia, México
  - Centro Potosino de Investigacion Medica S.C., San Luis Potosí City
- Netherlands (2):
  - Local Institution - 0335, Amsterdam, North Holland
  - Local Institution, Rotterdam
- New Zealand (4):
  - Auckland City Hospital, Auckland
  - Local Institution - 0271, Christchurch
  - Local Institution - 0268, Dunedin
  - Local Institution - 0269, Tauranga
- Norway (2):
  - Local Institution - 0213, Bergen
  - Local Institution - 0048, Oslo
- Peru (2):
  - Local Institution - 0179, Santiago de Surco, Lima region
  - Local Institution - 0385, Lima
- Poland (15):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Local Institution - 0414, Olsztyn, Warmian-Masurian Voivodeship
  - Local Institution - 0336, Biała Podlaska
  - Local Institution - 0120, Gdansk
  - Wojewodzkie Centrum Onkologii, Gdansk
  - Local Institution - 0377, Krakow
  - Local Institution - 0252, Krakow
  - Local Institution - 0373, Krakow
  - Instytut MSF Sp zoo, Lodz
  - Local Institution - 0118, Lublin
  - Local Institution - 0178, Poznan
  - Wojskowy Instytut Medyczny, Warsaw
  - Local Institution - 0328, Warsaw
  - Local Institution, Warsaw
  - Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw
- Portugal (3):
  - Local Institution - 0184, Lisbon
  - Local Institution - 0177, Lisbon
  - Local Institution - 0142, Porto
- FDI Clinical Research, San Juan, PR, Puerto Rico
- Romania (9):
  - Onco Clinic Consult SA, Craiova, Dolj
  - Local Institution - 0310, Bucharest, Sector 2
  - Institutul Oncologic Bucuresti IOB, Bucharest
  - Local Institution - 0127, Cluj-Napoca
  - Institutul Oncologic Prof. Dr. I. Chiricuta, Cluj-Napoca
  - Local Institution - 0189, Cluj-Napoca
  - Centrul de Oncologie Sf Nectarie, Craiova
  - Local Institution - 0133, Oradea
  - Sc Sigmedical Srl, Suceava
- Russia (4):
  - Local Institution - 0257, Krasnodar, Krasnodarskiy Kray
  - Local Institution - 0256, Krasnoyarsk
  - N.N. Blokhin National Medical Research Center of Oncology, Moscow
  - VitaMed LLC, Moscow
- South Korea (7):
  - Local Institution - 0389, Seongnam-si, Gyeonggi-do
  - Asan Medical Center, Seoul, Songpa-gu
  - National Cancer Center, Gyeonggi-do
  - Local Institution - 0221, Seongnam-si
  - Local Institution - 0206, Seoul
  - Local Institution - 0324, Seoul
  - Local Institution - 0207, Suwon
- Spain (32):
  - Local Institution - 0047, Donostia / San Sebastian, Guipuzcoa
  - Local Institution - 0287, Majadahonda, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Local Institution - 0122, A Coruña
  - Local Institution - 0382, A Coruña
  - Local Institution - 0173, Alicante
  - Catalan Institute of Badalona Hospital Germans Trias i Pujol ICO, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Local Institution - 0026, Barcelona
  - Local Institution - 0225, Barcelona
  - Local Institution, Barcelona
  - Local Institution - 0146, Burgos
  - Local Institution - 0144, Granada
  - Local Institution - 0273, Madrid
  - Local Institution - 0357, Madrid
  - Clinica Universidad de Navarra Madrid, Madrid
  - Local Institution - 0008, Madrid
  - Local Institution, Madrid
  - Local Institution - 0027, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Local Institution - 0192, Málaga
  - Local Institution, Santa Cruz de Tenerife
  - Local Institution - 0352, Santander
  - Local Institution - 0274, Seville
  - Local Institution - 0294, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario y Politecnico de La Fe, Valencia
- Sweden (3):
  - Local Institution, Gothenburg
  - Local Institution - 0036, Malmo
  - Local Institution, Umeå
- Switzerland (3):
  - Local Institution - 0119, Basel
  - Local Institution - 0403, Sankt Gallen
  - UniversitaetsSpital Zuerich - Dermatology, Zurich
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung
  - Local Institution - 0197, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital TPVGH, Taipei
- Local Institution - 0330, Ankara, Turkey (Türkiye)
- United Kingdom (10):
  - Local Institution - 0141, London, Greater London
  - University College Hospital, London, Greater London
  - Local Institution - 0272, London, Greater London
  - Local Institution - 0086, London, Greater London
  - The Christie Hospital, Manchester, Greater Manchester
  - Local Institution - 0195, Southampton, Hampshire
  - Local Institution - 0231, Maidstone, Kent
  - Local Institution - 0161, Northwood, Middlesex
  - Local Institution - 0299, Edinburgh, Scotland
  - Local Institution - 0259, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT03899155.html